CLINICAL TRIAL: NCT05303311
Title: Comparing the Analgesic Properties of Intrathecal Pethidine Plus Dexamethasone Versus Intrathecal Bupivacaine Alone for Distal Lower Extremity Orthopedic Surgeries: A Randomized Comparative Study.
Brief Title: Intrathecal Pethidine Plus Dexamethasone for Distal Lower Orthopedic Surgeries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Salwa Samir El Sherbeny, Lecturer of Anesthesia, Intensive Care and pain management, Faculty of Medicine, Zagazig University, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8035-7-11-2021
Record Dates: First submitted 2022-03-10; First posted 2022-03-31 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Meperidine; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine group (Active Comparator): Patients will be anesthetized by spinal anesthesia by intrathecal injection of 3 ml hyperbaric bupivacaine 0.5% alone.
  Interventions: Drug: Bupivacaine Hydrochloride
- pethidine plus dexamethasone group (Active Comparator): Patients will be anesthetized by spinal anesthesia by intrathecal injection of 1mg/kg preservative-free pethidine plus 4mg dexamethasone diluted to a volume of 3 ml with 0.9% sodium chloride
  Interventions: Drug: Pethidine plus Dexamethasone

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — intrathecal injection of bupivacaine alone
  Other Names: Heavy marcaine
  Arms: Bupivacaine group
Drug: Pethidine plus Dexamethasone — Intrathecal injection of pethidine plus dexamethasone
  Other Names: meperidine and decadron
  Arms: pethidine plus dexamethasone group

SUMMARY:
Bupivacaine is commonly used as a sole agent for spinal anesthesia unlike pethidine. Pethidine (meperidine) is a unique opioid. In addition to its analgesic activity, it also has significant local anesthetic activity. This property enables it to be used as the sole agent for spinal anesthesia

DETAILED DESCRIPTION:
pethidine compared favorably with bupivacaine as the sole anesthetic agent, providing excellent conditions for lower abdominal and pelvic surgery. Some studies showed that intrathecal pethidine has short motor recovery and prolonged postoperative analgesia in comparison to intrathecal bupivacaine. The side effects of pethidine in spinal anesthesia are pruritus nausea, vomiting and respiratory depression. A dose of 1mg/kg intrathecal pethidine provides surgical anesthesia .However, its effects are not widely available in recent studies.

Dexamethasone is used as an adjuvant to local anesthetic during spinal anesthesia and other techniques of regional anesthesia, it reduces pain and prolongs the duration of post-operative analgesia. It was shown that intrathecal dexamethasone reduces the complications of spinal anesthesia such as arterial hypotension, nausea, vomiting and shivering. The investigators suppose that addition of intrathecal dexamethasone to pethidine may be a better alternative to intrathecal bupivacaine during spinal anesthesia for lower extremity orthopedic surgery with better outcome and less side effects

ELIGIBILITY:
Inclusion Criteria:

* Patient acceptance.
* Patients scheduled for lower extremity orthopedic surgery
* Both sex
* Patient's age >18 years.
* Patients with American Society of Anaesthesia (ASA)physical status I, II.

Exclusion Criteria:

* Patient's age ≤18 years.
* Uncooperative patients and patients with psychological problems.
* Patients with contraindications to spinal anesthesia.
* Patients with contraindications to bupivacaine or dexamethasone or pethidine.
* Patients with ASA physical status III and IV.
* Morbid obesity (BMI >35).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
The Time of the first need for Rescue Analgesia | 24 hours postoperative
  the time from the end of the intrathecal injection of the study drugs to the first report of pain that reached NRS 4 as described by the patient.

SECONDARY OUTCOMES:
Intraoperative changes in the blood pressure measurements (The incidence of hypotension ) | duration of the procedure
  The incidence of hypotension "defined as the mean arterial blood pressure decreased by > 20 % from its value before intrathecal injection of the study drugs"
Intraoperative changes in the heart rate measurements (The incidence of bradycardia) | duration of the procedure
  bradycardia "defined as the reduction of heart rate by > 20% of the basal reading".
The onset of the sensory block | duration of the procedure
  The sensory level was checked using the pinprick technique every min for 10 min then at 2-min intervals until a constant block was obtained
The onset of the motor block | duration of the procedure
  The Motor Block was checked using Modified Bromage Score "Bromage 0 means full movement of the hip, knee, and ankle, Bromage 1 means loss of the ability to raise the leg against gravity but able to bend the knee and the ankle joints, Bromage 2 lost the ability to flex the hip and knee joints but preserved flexion of the ankle, Bromage 3 lost the ability to flex the hip, knee, and ankle joints but preserved movement of the toes, Bromage 4 indicates full paralysis of the legs". every min for 10 min then at 2-min intervals until a Bromage score 4 was obtained
The time of regression of sensory block to the 5th lumbar dermatome | Up to 12 hours postoperative
  The sensory level was checked using the pinprick technique every 15 min until sensations were gained back to the 5th lumbar dermatome
The time of regression of motor block to full motor function "Bromage score 0". | Up to 12 hours postoperative
  The Motor Block was checked using Modified Bromage Score every 15 min until full motor function was restored. "Bromage score 0"......
  Modified Bromage Score: "Bromage 0 means full movement of the hip, knee, and ankle, Bromage 1 means loss of the ability to raise the leg against gravity but able to bend the knee and the ankle joints, Bromage 2 lost the ability to flex the hip and knee joints but preserved flexion of the ankle, Bromage 3 lost the ability to flex the hip, knee, and ankle joints but preserved movement of the toes, Bromage 4 indicates full paralysis of the legs".
The incidence of perioperative adverse events | duration of the procedure and 24 hours postoperative
  Assess the frequency of perioperative nausea, vomiting, sedation, shivering, pruritis, and respiratory depression.

CONTACTS AND LOCATIONS:
Overall Officials: Salwa S ElSherbeny, Lecturer, Principal Investigator — Zagazig University
Locations (1):
- Faculty of Medicine , Zagazig University, Zagazig, Sharqia Province, Egypt